CLINICAL TRIAL: NCT01831518
Title: Evaluation of a Novel Method of Non-surface Electrocardiographic Mapping in Predicting Clinical, Structural and Neurohormonal Responses in Patients Undergoing Cardiac Resynchronization Therapy.
Brief Title: Predicting Response to CRT Using Body Surface ECG Mapping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tom Jackson (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); CardioInsight Technologies, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Tom Jackson, Clinical Research Fellow, Guy's and St Thomas' NHS Foundation Trust
Organization: Guy's and St Thomas' NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STHCIT1
Record Dates: First submitted 2013-04-04; First posted 2013-04-15 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure
Keywords: Heart Failure; Cardiac Resynchronization Therapy; ECG Imaging; Body Surface Mapping
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy; Cardiac Resynchronization Therapy Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CRT Eligible (Experimental): ACC/AHA/HRS/ESC guidelines for device-based therapy
  Interventions: Device: CRT Implant; Device: Body Surface ECG Mapping

INTERVENTIONS:
Device: CRT Implant
  Other Names: Cardiac Resynchronization; Biventricular Pacemaker
Device: Body Surface ECG Mapping
  Other Names: ECG Imaging

SUMMARY:
Cardiac resynchronization therapy (CRT) involves pacing the left and right side of the heart in order to improve the coordination of the contraction in patients with heart failure. Current selection criteria incorporate the severity of the symptoms, the mechanical function of the heart and the time it takes the electrical stimulation to spread over the left ventricle (as assessed on the standard 12 lead electrocardiogram-ECG). Unfortunately these criteria only seem to select approximately 70% of the patients who might respond to this invasive therapy. Body surface ECG mapping is a new technique that assesses the electrical activation of the heart in more detail than the standard ECG. This study aims to determine whether this new technology may aid current selection criteria in predicting response to CRT.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Fulfils established clinical criteria for CRT implantation (with or without a defibrillator)
* NYHA Class III-IV Heart Failure (or NYHA II with NYHA III/IV symptoms in the preceding 12 months)
* LVEF <35% (Calculated using echocardiography or Cardiac MR) at the time of implantation
* QRS duration > 130ms
* Optimal Tolerated Medical Therapy for Heart Failure

Exclusion Criteria:

* Severe, life threatening non cardiac disease
* Active malignant disease and recent (<5 years) malignant disease
* Prior Heart Transplant
* Recent history of unstable angina, acute coronary syndrome or myocardial infarction within three months of enrolment into the study
* Pregnancy
* Failure to participate in consent process
* Atrial Fibrillation
* Conventional pacemaker in situ
* Heart Failure requiring constant intravenous therapy including diuretics and/or inotropes
* Recent revascularisation procedure i.e. coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI) within the last three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Change in distance travelled during six-minute walk test (6MWT) | Baseline and 6 months
Echocardiographic: signs of LV reverse remodelling | Baseline and 6 months
  Increase by >5% in left ventricular ejection fraction with an associated decrease in LV end-diastolic (LVEDV) and end-systolic (LVESV) volumes

SECONDARY OUTCOMES:
Symptoms | Baseline and 6 months
  Change in symptoms severity assessed by Minnesota Living With Heart Failure Questionnaire (MLHFQ)
Neurohormonal status | Baseline and 6 Months
  Change in neurohormonal activation assessed by brain-natriuretic peptide (BNP)
Pacing | 6 months
  Atrial and ventricular arrhythmic burden, percentage of bi-ventricular pacing

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - The Royal Brompton and Harefield NHS Foundation Trust, London

REFERENCES:
- [Derived] Jackson T, Claridge S, Behar J, Sieniewicz B, Gould J, Porter B, Sidhu B, Yao C, Lee A, Niederer S, Rinaldi CA. Differential effect with septal and apical RV pacing on ventricular activation in patients with left bundle branch block assessed by non-invasive electrical imaging and in silico modelling. J Interv Card Electrophysiol. 2020 Jan;57(1):115-123. doi: 10.1007/s10840-019-00567-2. Epub 2019 Jun 14. PMID 31201592